CLINICAL TRIAL: NCT01945099
Title: Acceleration of Insulin Action by Hyaluronidase During Closed-Loop Therapy
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 1307012334
Record Dates: First submitted 2013-07-17; First posted 2013-09-18 (Estimated); Last update posted 2022-05-24 (Actual); Status verified 2022-05

CONDITIONS: Type 1 Diabetes
Keywords: diabetes, insulin,post prandial, closed loop, artificial pancreas, hyperglycemia
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus; Hyperglycemia | interventions — Hyaluronoglucosaminidase

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- ePID closed loop system without hyaluronidase (Active Comparator): Hyaluronidase will not be given while subject uses ePID closed loop system
  Interventions: Device: ePID closed loop system
- ePID closed loop system with hyaluronidase at infusion site (Experimental): Hyaluronidase will be injected at insulin pump infusion site prior to the time that subject uses ePID closed loop system
  Interventions: Device: ePID closed loop system; Drug: hyaluronidase
- ePID closed loop system with hyaluronidase co-formulation (Experimental): Hyaluronidase-insulin co-formulation will be used in study pump while subject uses ePID closed loop system
  Interventions: Device: ePID closed loop system; Drug: Lispro-PH20

INTERVENTIONS:
Device: ePID closed loop system — Insulin pump controlled by closed loop unit and algorithm
Drug: hyaluronidase
  Other Names: rHuPH20
  Arms: ePID closed loop system with hyaluronidase at infusion site
Drug: Lispro-PH20
  Other Names: insulin-hyaluronidase co-formulation
  Arms: ePID closed loop system with hyaluronidase co-formulation

SUMMARY:
"Closed loop artificial pancreas" systems have been under development for the control of blood sugars in those living with diabetes. These systems consist of a continuous glucose sensor, which sends a signal to a computer program that automatically determines how much insulin to give. The computer program then tells an insulin pump to deliver the insulin. While such systems have been tested under a number of conditions, post-meal blood sugars are difficult to control. Specifically, we will be looking to see if using hyaluronidase improves the ability of the closed loop artificial pancreas to better respond to meal related highs and lows.

DETAILED DESCRIPTION:
To investigate the effect of rHuPH20, an adjuvant that accelerates the dispersion and absorption of subcutaneously injected or infused drugs, on mitigating post-prandial blood glucose excursions when injected separately or co-formulated with insulin during closed-loop therapy for youth and young adults with type 1 diabetes. Closed-loop control will be achieved using external subcutaneous real-time continuous glucose monitoring and continuous subcutaneous insulin infusion along with a computerized algorithm to link these two processes.

Specific Aim 1: To examine whether co-formulation rHuPH20 with analog insulin (INS-PH20)or, alternately, pre-administration of rHuPH20 (PH20-preRx) at the time of infusion set placement prior to initiation of closed-loop (CL) insulin delivery will reduce peak-postprandial glucose concentrations and total glucose area under the curve of the meal excursions in short term inpatient experiments.

Specific Aim 2: To investigate whether accelerated insulin absorption by rHuPH20, delivered as described above, will also result in a reduction of late-post-prandial hyperinsulinemia and late post-prandial hypoglycemia during CL insulin delivery.

Specific Aim 3: To compare the insulin accelerator effect of INS-PH20 to that of PH20-preRx, based on post prandial glucose excursions during closed-loop therapy

We hypothesize that; utilization of PH20 either as a separate injection (PH20-preRx) or in a co-formulation with insulin (INS-PH20) during CL therapy will reduce peak-postprandial glucose concentrations and total glucose under the curve of the meal excursion as compared to CL control without any intervention, and we propose that the use of PH20-preRx and INS-PH20 will be well tolerated when delivered in youth and young adults in a closed-loop setting.

ELIGIBILITY:
Inclusion Criteria:

1. age 12-40 years
2. clinical diagnosis of T1D based on ADA criteria or presence of DKA at diagnosis (formal antibody and/or genetic testing will not be required)
3. duration of T1D ≥ 1 year
4. HbA1c ≤ 9 %
5. Treated with CSII for at least 3 months
6. Body weight > 37 kg (to accommodate phlebotomy)
7. Normal hematocrit
8. Normal creatinine
9. Not pregnant or lactating, and for female subjects of reproductive potential, are abstinent or are consistently using barrier or hormonal methods of contraception

Exclusion Criteria:

1. Insulin resistant (defined as requiring > 2 units/kg/day at time of study enrollment
2. Previous allergic reaction to PH20
3. Inability to comprehend written or spoken English
4. Presence of any medical or psychiatric disorder that may interfere with subject safety or study conduct
5. Use of any medications (besides insulin) known to affect blood glucose levels, including oral or other systemic glucocorticoid therapy. Inhaled, intranasal, or rectal corticosteroid use is allowed along as not given within 4 weeks of admission to the HRU. Use of topical glucocorticoids is allowable as long as affected skin area does not overlap with study device sites. Subjects using herbal supplements will be excluded, due to the unknown effects of these supplements on glucose control
6. Use of furosemide, benzodiazepines or phenytoin during the study
7. History of poor wound healing, heat sensitivity, or diminished skin integrity.
8. History of hypoglycemic seizure within last 3 months
9. Anemic (low hematocrit), or evidence of renal insufficiency (elevated serum creatinine)
10. Female subjects who are pregnant, lactating, or unwilling to be tested for pregnancy
11. Subjects unable to give consent / permission / assent

Ages: 12 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 13 (Actual)
Dates: Start 2013-09; Primary Completion 2015-12 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Peak post-prandial venous glucose levels obtained after breakfast, lunch, and dinner between CL alone and CL+PH20preRx and CL+INS-PH20 | during each admission for 3 consecutive study visit days
  Peak post-prandial plasma glucose excursions (mg/dL) after breakfast, lunch, and dinner on days #2, #3 and #4. One day with hylauronidase pre-treated insulin infusion site site, other day with hyaluronidase-rapid acting insulin co-formulation infusion and control day with rapid acting insulin only.

SECONDARY OUTCOMES:
Peak post-prandial insulin levels following meals | during each admission for 3 consecutive study visit days

OTHER OUTCOMES:
Area Under Curve meal-related insulin excursion following meals | during each admission for 3 of the study days

CONTACTS AND LOCATIONS:
Overall Officials: Eda Cengiz, MD, MHS, Principal Investigator — Yale University
Locations (1):
- Yale University School of Medicine, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No